CLINICAL TRIAL: NCT02723448
Title: A Pilot Study of Aclarubicin for the Treatment of Retinal Vasculopathy With Cerebral Leukodystrophy (RVCL)
Brief Title: Aclarubicin for the Treatment of Retinal Vasculopathy With Cerebral Leukodystrophy
Acronym: RVCL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, John P. Atkinson, MD, Professor of Medicine, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATK2016001
Record Dates: First submitted 2016-03-02; First posted 2016-03-30 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Vasculopathy, Retinal, With Cerebral Leukodystrophy; Cerebroretinal Vasculopathy, Hereditary
MeSH Terms: conditions — Vasculopathy, Retinal, With Cerebral Leukodystrophy | interventions — Aclarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Study (Other): Aclarubicin (6 mg/m²) will be administered intravenously through a central venous access device over 1 hour for four consecutive days (Days 2-5) of each 28 day cycle to each participant [Retinal Vasculopathy with Cerebral Leukodystrophy (RVCL) patients]. There is no maximum number of cycles.
  Interventions: Drug: aclarubicin

INTERVENTIONS:
Drug: aclarubicin — Aclarubicin (3 mg/m²) will be administered intravenously through a central venous access device over 1 hour for four consecutive days per 28 day cycle. There is no maximum number of cycles.
  Other Names: aclacinomycin-A (HCl)

SUMMARY:
The goal of the investigator is to utilize Aclarubicin to treat patients with Retinal Vasculopathy with Cerebral Leukodystrophy (RVCL), a rare and devastating genetic disease with no available specific treatment. RVCL results from a mutation in the tail end of the TREX1 (Three Prime Repair Exonuclease 1) gene, a major deoxyribonucleic acid (DNA) repair enzyme. The RVCL-specific mutations cause expression of a truncated and mislocalized protein. RVCL is an inherited disorder whose symptoms begin at middle age and initially predominantly affects the eye and brain. Because it is an 'autosomal dominant' disease, it strikes both males and females equally. A person with RVCL has a 50-50 chance of transmitting the gene to each child.

The investigator's published studies demonstrated in a mouse model for RVCL and in vitro studies with patients' cells that defects were corrected by use of Aclarubicin, an anthracycline antibiotic often used to treat cancer. Thus, there is a strong rationale for conducting a clinical trial of aclarubicin in patients with RVCL.

The dosage to be initially administered to RVCL patients initially will be < 10% of that typically used in cancer therapeutics and will be given monthly on four consecutive days for six months. Patients will undergo assessments every six months to determine disease response. Patients that do not have clear objective response may be dose escalated by 1 dose level with permission of the principal investigator permitting the patient has not previously experienced any toxicities requiring dose modifications. We will evaluate the safety and clinical efficacy of Aclarubicin for the treatment of RVCL and evaluate its effects on cellular function. This work will generate the first clinical research data on the investigational product's utility in treating RVCL.

Patients are followed for at least 2 years upon completion of Aclarubicin administration completion. We are not longer administering the drug, but are in the post-drug follow up arm of the study.

DETAILED DESCRIPTION:
Retinal vasculopathy with cerebral leukodystrophy (RVCL) is a very rare and uniformly fatal genetic condition that affects the microvasculature. Symptoms begin in adulthood (usually in the 40s) and include loss of vision, mini-strokes, and dementia. RVCL includes three conditions which were previously thought to be distinct: hereditary endotheliopathy, retinopathy, nephropathy, and stroke (HERNS); cerebroretinal vasculopathy (CRV); and hereditary vascular retinopathy (HVR). RVCL is inherited in an autosomal dominant manner and is caused by carboxyl (C)-terminal heterozygous frameshift (fs) mutations in TREX1 (Three Prime Repair Exonuclease 1). There is no treatment for RVCL, only symptomatic management.

TREX1 is an endoplasmic reticulum (ER)-associated (i.e., intracellular) enzyme that, in addition to its DNA repair activities, may regulate sugar metabolism in the ER. TREX1 mutations have also been associated with several autoimmune and autoinflammatory diseases. In RVCL, fs mutations of TREX1 result in C-terminal truncation and this dysregulates the oligosaccharyltransferase (OST) complex leading to free glycan release from dolichol carriers. In mouse models and in patient-derived cells, inhibiting OST with aclarubicin may correct glycan and immune defects associated with fs mutations of TREX1 (Hasan, M. et al., Immunity 43: 1-12, 2015).

Aclarubicin (aka aclacinomycin, aclacinomycin-A) is an anthracycline antibiotic isolated from Streptomyces galilaeus cultures. Aclarubicin has been shown to have a broad spectrum of anti-tumor activity. Aclarubicin was utilized for treatment of various cancers in Phase 1 and 2 studies in the United States of American (USA) in the 1980's and 1990's. While no longer clinically employed in the USA, it is commonly used in China and Japan, often as part of a combination drug therapy program for certain malignancies.

Aclarubicin is typically administered over 3-5 consecutive days, however, alternative schedules such as weekly or monthly have been evaluated. In solid tumors, the maximum tolerated dose (MTD) of 4-day dosing was 30 mg/m2/day; marrow suppression was dose limiting, otherwise the regimen was well tolerated. Additionally, a Phase II study in acute myeloblastic leukemia was conducted using 100mg/m2 per day for three days and repeated at days 14-16 if marrow hypoplasia was not produced. Toxic effects of this regimen included severe neutropenia, nasea/vomiting, and diarrhea. No changes were noted in left ventricular ejection fraction or no cardiac symptoms developed.

RVCL is caused by fs mutations in the C-terminus of TREX1 resulting in low-grade free glycan release, immune activation, and possibly autoantibody production due in part to dysregulation of the OST complex. Inhibiting OST with aclarubicin corrects these glycan and immune defects in mouse models and in patient-derived cells. Thus, inhibiting OST with aclarubicin might be a therapeutic option for patients with RVCL.

Given the poor prognosis of RVCL, the lack of treatment options, and the pre-clinical data on OST inhibition by aclarubicin in mice, there is strong rationale for conducting a clinical trial of aclarubicin in patients with RVCL.

In this pilot study, aclarubicin will be administered initially at ~ 20% of the single-agent maximum tolerated dose (MTD) in oncology studies. Assessments will be made every six months as to objectives of the study. Patients that do not have clear objective response may have their dose level increased with permission of the principal investigator permitting the patient has not previously experienced any toxicities requiring dose modifications. A patient who has clear objective progression at any time may also have their dose escalated as long as they have completed 1 full cycle at their current dose level. Maximum dose level will be 24 mg/m2/day. The aim of aclarubicin administration in RVCL is not to induce apoptosis, as in oncology studies, but rather to modulate intracellular functions and, thus, a reduced dose will be utilized.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of Retinal Vasculopathy with Cerebral Leukodystrophy (RVCL)
2. At least 18 years of age at the time of study registration
3. Normal hematologic function defined as: WBC (white blood cell count) > 4 x10⁹/L, ANC (absolute neutrophil count) ( >1.5 x 10⁹/L and Platelets > 100 x10⁹/L
4. Females of childbearing potential (FCBP) must agree to refrain from becoming pregnant while on study drug and for 3 months after discontinuation from study drug, and must agree to use adequate contraception including hormonal contraception, (i.e. birth control pills, etc), barrier method contraception (i.e. condoms), or abstinence during that time frame.
5. Able to understand and willing to sign an IRB (Institutional Review Board) approved written informed consent document (or that of legally authorized representative, if applicable)

Exclusion Criteria:

1. Acute bacterial, fungal, or viral infection
2. Known human immunodeficiency virus (HIV) or active hepatitis B or C virus infection
3. Pregnant and/or breastfeeding
4. Cardiovascular disease including: congestive heart failure [left ventricular ejection fraction (LVEF) < 55%] at screening; electrocardiogram (EKG) evidence of acute ischemia or medically significant conduction system abnormalities; or unstable arrhythmia or angina
5. Cumulative prior anthracycline dose of 300 mg/m²
6. Known hypersensitivity to one or more of the study agents
7. Currently receiving or has received any investigational drugs within the 14 days prior to the first dose of study drug
8. Currently receiving or has received any immunosuppressants within the 14 days prior to the first dose of study drug

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Change in Lesion Pattern on Fluid-Attenuated Inversion Recovery (FLAIR) Magnetic Resonance Imaging (MRI) in Retinal Vasculopathy Cerebral Leukodystrophy (RVCL) patients | Change from baseline at six months
  Volume increase in lesions on FLAIR MRI between baseline and six months is assessed

CONTACTS AND LOCATIONS:
Overall Officials: John P Atkinson, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared among the principal investigator and the sub-investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data is currently being shared among the principal investigator and the subinvestigators
Access Criteria: IPD is available on REDCap or as provided by principal investigator

REFERENCES:
- [Background] Hasan M, Fermaintt CS, Gao N, Sakai T, Miyazaki T, Jiang S, Li QZ, Atkinson JP, Morse HC 3rd, Lehrman MA, Yan N. Cytosolic Nuclease TREX1 Regulates Oligosaccharyltransferase Activity Independent of Nuclease Activity to Suppress Immune Activation. Immunity. 2015 Sep 15;43(3):463-74. doi: 10.1016/j.immuni.2015.07.022. Epub 2015 Aug 25. PMID 26320659
- [Background] Kavanagh D, Spitzer D, Kothari PH, Shaikh A, Liszewski MK, Richards A, Atkinson JP. New roles for the major human 3'-5' exonuclease TREX1 in human disease. Cell Cycle. 2008 Jun 15;7(12):1718-25. doi: 10.4161/cc.7.12.6162. Epub 2008 Jun 16. PMID 18583934
- [Background] Karanes C, Young JD, Samson MK, Smith LB, Franco LA, Baker LH. Phase I trial of aclacinomycin-A. A clinical and pharmacokinetic study. Invest New Drugs. 1983;1(2):173-9. doi: 10.1007/BF00172077. PMID 6590531
- [Background] Kerpel-Fronius S, Gyergyay F, Hindy I, Decker A, Sawinsky I, Faller K, Mechl Z, Nekulova M, Kolaric K, Tomek R, et al. Phase I-II trial of aclacinomycin A given in a four-consecutive-day schedule to patients with solid tumours. A South-East European Oncology Group (SEEOG) Study. Oncology. 1987;44(3):159-63. doi: 10.1159/000226469. PMID 3474571
- [Background] Case DC Jr, Ervin TJ, Boyd MA, Bove LG, Sonneborn HL, Paul SD. Phase II study of aclarubicin in acute myeloblastic leukemia. Am J Clin Oncol. 1987 Dec;10(6):523-6. doi: 10.1097/00000421-198712000-00014. PMID 3479891
- [Background] Stam AH, Kothari PH, Shaikh A, Gschwendter A, Jen JC, Hodgkinson S, Hardy TA, Hayes M, Kempster PA, Kotschet KE, Bajema IM, van Duinen SG, Maat-Schieman MLC, de Jong PTVM, de Smet MD, de Wolff-Rouendaal D, Dijkman G, Pelzer N, Kolar GR, Schmidt RE, Lacey J, Joseph D, Fintak DR, Grand MG, Brunt EM, Liapis H, Hajj-Ali RA, Kruit MC, van Buchem MA, Dichgans M, Frants RR, van den Maagdenberg AMJM, Haan J, Baloh RW, Atkinson JP, Terwindt GM, Ferrari MD. Retinal vasculopathy with cerebral leukoencephalopathy and systemic manifestations. Brain. 2016 Nov 1;139(11):2909-2922. doi: 10.1093/brain/aww217. PMID 27604306